CLINICAL TRIAL: NCT03304925
Title: CoolSculpting the Flanks
Acronym: CSI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA17-002
Record Dates: First submitted 2017-10-03; First posted 2017-10-09 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Body Fat Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Fat Reduction (Experimental): The treatments are designed to see if the fat can be reduced in the flanks with a new applicator design.
  Interventions: Device: The ZELTIQ System

INTERVENTIONS:
Device: The ZELTIQ System — The CoolSculpting machine will be used to perform the treatments.

SUMMARY:
Evaluate the safety and efficacy of non-invasive subcutaneous fat layer reduction in the flanks.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects > 22 years of age and < 65 years of age.
* Subject has clearly visible fat on the flanks, which in the investigator's opinion, may benefit from the treatment.
* No weight change exceeding 5% of body weight in the preceding month.
* Subject with body mass index (BMI) up to 30. BMI is defined as weight in pounds multiplied by 703 divided by the square of the height in inches.
* Subject agrees to maintain his/her weight (i.e., within 5%) by not making any major changes in their diet or exercise routine during the course of the study.
* Subject has read and signed the study written informed consent form.

Exclusion Criteria

* Subject has had a surgical procedure(s) in the area of intended treatment.
* Subject has had an invasive fat reduction procedure (e.g., liposuction, mesotherapy) in the area of intended treatment.
* Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 12 months.
* Subject needs to administer, or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
* Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
* Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
* Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
* Subject is taking or has taken diet pills or supplements within the past month.
* Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
* Subject has an active implanted device such as a pacemaker, defibrillator, or drug delivery system
* Subject is pregnant or intending to become pregnant during the study period (in the next 8 months).
* Subject is lactating or has been lactating in the past 6 months.
* Subject has a history of hernia in the areas to be treated.
* Subject is unable or unwilling to comply with the study requirements.
* Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2017-10-25 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Safety endpoint in relation to adverse events | Final post treatment visit
  Measurement of device- or procedure-related adverse events. It is expected there will be zero UADEs
Effectiveness endpoint gauged by reduction in fat layer thickness | Final post-treatment visit
  Reduction in fat layer thickness as measured by ultrasound at the final post-treatment visit.

SECONDARY OUTCOMES:
Subject survey | Final post-treatment visit
  Subject survey as assessed by questionnaire administered at the final post-treatment visit.
Photo review | Final post-treatment visit
  Correct identification of pre-treatment vs. final post-treatment visit images by two out of three blinded independent reviewers.

CONTACTS AND LOCATIONS:
Overall Officials: Kerrie Jiang, NP, Study Director — Zeltiq Aesthetics
Locations (7):
- United States (7):
  - Innovation Research Center, Pleasanton, California
  - Laser & Skin Surgery Center of Northern California, Sacramento, California
  - SkinCare Physicians of Chestnut Hill, Chestnut Hill, Massachusetts
  - Zel Skin & Laser Specialist, Edina, Minnesota
  - Laser & Skin Surgery Center of New York, New York, New York
  - Brian S. Biesman, MD, Nashville, Tennessee
  - EpiCenter Skincare and Laser Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No